CLINICAL TRIAL: NCT02957422
Title: Dairy Intake and Cerebral Antioxidant Defense in Aging: a Dietary Intervention Study
Brief Title: Milk Intervention Study for Brain Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00140131
Record Dates: First submitted 2016-11-04; First posted 2016-11-07 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Brain Aging
Keywords: milk; brain aging; antioxidant; glutathione; dietary intervention; brain imaging
MeSH Terms: interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention (Experimental): Participants will receive dietary intervention. Participants will be taking 3 servings of dairy/day.
  Interventions: Dietary Supplement: 1% Milk
- Control (Active Comparator): Participants will receive no additional intervention. Participants will continue on their regular diet, which includes ≤1.5 dairy serving/day.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: 1% Milk — 1.5 gallons of 1% milk will be delivered to the participant's home weekly. Participants will be asked to drink 3 cups per day for 3 months.
  Arms: Dietary intervention
Dietary Supplement: Control — Participants will continue on their regular low dairy diet of ≤1.5 dairy serving/day.
  Arms: Control

SUMMARY:
The purpose of this study is to learn if increased dairy food consumption helps brain health in older adults by protecting nerve cells from damage.

DETAILED DESCRIPTION:
Eating more dairy foods may improve brain health as people age by increasing the brain's natural defenses to protect nerve cells against chemical stress. Researchers think there may be a relationship between the brain's natural defense system and the amount of dairy food intake. Strengthening these defenses could provide beneficial protection to the brain against neurodegenerative age-related diseases and cognitive decline.

Glutathione (GSH) is a metabolite in the human brain protective system. It plays a key role in protecting cells against oxidative stress, which is one of the major processes contributing to aging and neurodegeneration. Preliminary findings suggest that there may be a correlation between dairy food intake and GSH levels in the aging brain. Magnetic Resonance Spectroscopy (MRS) measures chemicals in the brain. It is a noninvasive measure of the effects of dairy food intake on the major protective metabolite levels in the living human brain in aging.

This study involves using an MRI with special MRS scans to see if adequate dairy food intake may aid in enhancing cerebral protective capacity to fight against age-related disease and cognitive decline in the brain.

Participants will be asked to make a total of six visits to the research site. Participation will last about 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with no concomitant diseases which could interfere with the study
* Low dairy consumption (≤ 1.5 dairy serving/day)
* Mini-Mental State Exam (MMSE) ≥ 24
* body mass index (BMI) range: 18.5 - 35 kg/m2

Exclusion Criteria:

* Presence of any central neurological diseases or prior major head trauma with loss of consciousness
* Presence of an active unstable and life-threatening systemic illness (e.g., cancer)
* Presence of major psychiatric disorders within the past 3 years including depression, anxiety, and alcohol or drug abuse
* Presence of diabetes mellitus, metabolic syndrome or uncontrolled hypertension
* Use of psychoactive and investigational medications
* Subjects with MRI contraindications such as pacemaker, aneurysm clips, artificial heart valves, metal fragments, foreign objects or claustrophobia.
* Pregnancy
* Special diet regimens such as lactose free or vegan

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Change in Glutathione (GSH) levels | Change from Baseline to Month 3
  GSH levels are measured in frontal and parietal regions of the brain using our multiple quantum filtered chemical shift imaging (MQ CSI) technique with a 3 T clinical scanner.

CONTACTS AND LOCATIONS:
Overall Officials: In-Young Choi, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi IY, Taylor MK, Lee P, Alhayek SA, Bechtel M, Hamilton-Reeves J, Spaeth K, Adany P, Sullivan DK. Milk intake enhances cerebral antioxidant (glutathione) concentration in older adults: A randomized controlled intervention study. Front Nutr. 2022 Aug 15;9:811650. doi: 10.3389/fnut.2022.811650. eCollection 2022. PMID 36046132